CLINICAL TRIAL: NCT03948815
Title: Room 4 Birth - An Adaptable Birthing Room and the Effect on Labour and Birth: A Randomised Controlled Trial
Brief Title: Room 4 Birth - An Adaptable Birthing Room and the Effect on Labour and Birth
Acronym: R4B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Collaborators: Chalmers University of Technology (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Room 4 Birth - Swe
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Child Birth
Keywords: Birthing room; labour; randomised controlled trial

STUDY DESIGN:
Intervention Model Description: Decreased stress, increased parasympathisuc, increased physiological oxytocin promotes a normal healthy Labour and birth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention room (Experimental): An adaptable, person-centered, birthing room that is specially designed.
  Interventions: Other: interventional birthing room
- Control room (Other): A regular standard birthing room
  Interventions: Other: interventional birthing room

INTERVENTIONS:
Other: interventional birthing room — The design of the room is based on scientific evidence on the healthcare environment in general, and on a systematic review on the effect of birthing rooms published by the investigators, and interviews with women early after birth in Sweden. The room has a large birthing pool, several lighting options with dimming function, 40 mm suspended sound absorber in the ceiling, media installation covering two walls, which offers a choice of six different programmed nature scenes with light, sound effect and Music.

SUMMARY:
Healthcare Environment influences health outcomes. The effects of physical aspects of the birthing room on maternal and neonatal outcomes is insufficiently studied. This study will measure and compare effects and experiences of two types of birthing rooms.

DETAILED DESCRIPTION:
Healthcare Environment influences health outcomes. The effects of physical aspects of the birthing room on maternal and neonatal outcomes is insufficiently studied. This RCT project measures and compares effects and experiences of two types of birthing rooms at one Labour ward in Sweden. A qualitative ethnografic studu will assess how women interact with the birthing rooms and its physical objects.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* Robson 1 classified, i.e. nulliparous, single Pregnancy >37 weeks, cephalic presentation, sponatanous Labour start
* speak, understand Swedish, English, arabic or somali or have an interpreter present
* Active phase of Labour: 2 of these 3 criteria fulfilled: sponatanous rupture of membranes, 2-3 painful contractions in 10 minutes; cervix dilated >3-4 cm or effaced and open >1cm

Exclusion Criteria:

* induced Labour
* planned caesarean section
* multiple gestation
* lack of informed written consent
* not Speaking Swedish, Egmnlish, Arabic or Somali

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1268 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of four variables - Use of oxytocin (Y/N); Spontaneous vaginal birth (Y/N); Normal postpartum haemorrhage (Y/N); Self-rated childbirth experience | within 2 hours after birth
  Use of oxytocin for augmentation of Labour, Spontaneous vaginal birth, normal Postpartum haemorrhage, Childbirth experience

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldkuhl L, Tistad M, Gyllensten H, Berg M. Implementing a new birthing room design: a qualitative study with a care provider perspective. BMC Health Serv Res. 2023 Oct 19;23(1):1122. doi: 10.1186/s12913-023-10051-3. PMID 37858103
- [Derived] Berg M, Goldkuhl L, Nilsson C, Wijk H, Gyllensten H, Lindahl G, Uvnas Moberg K, Begley C. Room4Birth - the effect of an adaptable birthing room on labour and birth outcomes for nulliparous women at term with spontaneous labour start: study protocol for a randomised controlled superiority trial in Sweden. Trials. 2019 Nov 19;20(1):629. doi: 10.1186/s13063-019-3765-x. PMID 31744523